CLINICAL TRIAL: NCT04108871
Title: Randomized-controlled Trial: Whether Transperineal Prostate Biopsy Under Local-anaesthesia Using a Transperineal-access System is Non-inferior to Standard Transrectal Biopsy to Detect Prostate Cancer in Biopsy-naïve Men
Brief Title: Whether Transperineal Prostate Biopsy Under Local-anaesthesia Using a Transperineal-access System is Non-inferior to Standard Transrectal Biopsy to Detect Prostate Cancer in Biopsy-naïve Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wayne Lam, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UW18-392
Record Dates: First submitted 2019-05-14; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer; Prostatic Hyperplasia
Keywords: Biopsy; Transperineal Prostate Biopsy; Prostate Cancer Detection; Transrectal Prostate Biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transperineal Prostate Biopsy (Experimental): The biopsy needed is inserted to the prostate through the perineal skin, with the assistance of an access system device known as PrecisionPoint. It utilises a single access needle cannula mounted directly on to the ultrasound probe, which acts as an access point traversing through the perineal skin. 4 - 5 cores are obtained from the anterior, mid and posterior zone of each side of the prostate.
  Interventions: Procedure: Prostate Biopsy
- Transrectal Prostate Biopsy (Active Comparator): The biopsy needle penetrates through the bowel (rectum) to the prostate to obtain 12 cores of prostate tissues from the lateral and medial base, midzone and apex of each side of the prostate (1 core each).
  Interventions: Procedure: Prostate Biopsy

INTERVENTIONS:
Procedure: Prostate Biopsy — Samples of tissue are removed from the prostate for histopathological diagnosis of prostate cancer through the use of a needle with the assistance of transrectal ultrasound.

SUMMARY:
Tranperineal prostate biopsy(TPB) and Transrectal prostate biopsy(TRUSB) are now both routine diagnosis methods of prostate cancer in Queen Mary Hospital. The TRUSB has been the most common way to sample prostate tissue for decades. The TPB has been employed as one of our routine diagnosis methods in early 2018. The aim of this study is to evaluate whether Tranperineal prostate biopsy using a noval transperineal access system under local anaesthesia is non-inferior to standard 12-cores Transrectal prostate biopsy in detecting prostate cancer (PCa), in patients with clinical suspicion of PCa with no prior prostate biopsy.

DETAILED DESCRIPTION:
The incidence of prostate cancer (PCa) has increased considerably in recent years [1, 2]. The reported lifetime risk for men in Hong Kong to be diagnosed with PCa is 1 in 31 before the age of 75, and is currently the third commonest cancer Hong Kong men according to the Hong Kong Cancer Registry [3]. This highlights the importance of thorough and fundamentally a safe investigation technique to correctly identify patients with PCa. Such test should be able to sensitively detect PCa, and provide early diagnosis. Critically, such test is required to provide accurate disease risk stratification, which is absolutely crucial in guiding level of appropriate treatment is necessary in patients diagnosed with PCa.

According to recommendations from the National Institute for Health and Care Excellence (NICE) guidelines, current standard clinical practice considers histological diagnosis of PCa a necessity in majority of patients presented with localized disease who are eligible for treatment [4]. This, alongside with prostate specific antigen (PSA) level, digital rectal examination (DRE) findings, and increasingly the use of multi-parametric MRI (mpMRI) imaging, collectively allows risk stratification of PCa.

The current pathway to obtain prostate tissue for histological diagnosis of CaP is by transrectal ultrasound-guided systematic biopsy (TRUSB) of the prostate, usually following the detection of a raised serum PSA level and/or suspicious rectal examination findings. TRUSB has been the standard prostate tissue sampling technique for men suspected with PCa for over 30 years. It is an office-based procedure carried out under local anaesthesia (LA), with 10 to 12 biopsy cores directed towards the lateral peripheral zones of the prostate thought to harbour majority of cancers [7]. However, there are still various well-known cancer detection limitations and patient safety problems associated with TRUSB.

Firstly, a very significant portion of tumours are being missed with the TRUSB technique [8]. It has been well- known that over 30% of patients with low risk PCa on TRUSB have been found to harbour clinically significant PCa [9]. Many of these tumours missed on TRUSB are located in the anterior and apical regions of the prostate, which TRUSB is difficult to access, in particular in patients with a large prostate volume

Secondly, TRUSB requires the biopsy needle to penetrate through the bowel (rectum). This results in high risk of developing sepsis following biopsy, despite all patients undergoing the procedure being started on antibiotics prophylactically. This is a serious complication which can potentially be life-threatening. Our previous study has already demonstrated a high prevalence of fluoroquinolone-resistant and ESBL-producing rectal flora in our local population in Hong Kong [10]. The risk of developing post-biopsy sepsis in Hong Kong is high.

Transperineal prostate biopsy (TPB) has been developed to provide a more comprehensive biopsy method to improve cancer detection rate by directing biopsy cores through the perineal skin. Theoretically, TPB enables access to sample the entire prostate, in particular the anterior and apical regions which are not easily accessible through the standard TRUSB method. By sampling the prostate using biopsy needles directly inserted through the perineal skin rather than bowel, the risk of sepsis is reduced. However, this technique requires multiple needles traversing through the perineum, and requires to be carried out under general anaesthesia (GA). Another disadvantage is a stabilising stepping unit is required to provide a consistent alignment of the ultrasound probe against the prostate in order to carry out the biopsies. Such stabilising stepping units are costly.

A novel but simple transperineal access system device known as PrecisionPoint (Perineologic, Cumberland, MD, USA) has been developed to tackle the aforementioned limitations of TPB. This revolutionary device utilises a single access needle cannula mounted directly on to the ultrasound probe, which acts as an access point traversing through the perineal skin. This design minimises the number of needle punctures through the skin, enabling TPB to be carried out under LA. A stabilising stepping unit is not required with this technique. The device has gained the United States Food and Drug Administration (FDA) approval [11], and results from small contemporary series have already been published with very promising results in terms of cancer detection rate and safety [12].

TRUSB has a poor cancer detection rate and is associated with potentially fatal septic risk. TPB, if able to be carried out under LA as an office-based procedure, can potentially provide a better cancer detection rate with significantly reduced sepsis risk. It has fundamentally a very high potential to become the new gold standard in obtaining prostate tissue for histological diagnosis of PCa.

With an increasing number of men in Hong Kong with elevated serum PSA suspicion of PCa needing prostate biopsy, it is fundamental to carry out a study to determine the most effective, safe and tolerable prostate biopsy technique which fits with the clinical practice in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Serum PSA larger or equal to 20ng/mL
* Suspected tumour clinical stage T2 on DRE
* No previous history of prostate biopsy
* Medically fit to undergo procedures according to study protocol

Exclusion Criteria:

* Patients who are unable to provide written informed consent
* Known history of prostate cancer
* Contraindication to prostate biopsy
* Had pre-biopsy mpMRI
* Rectal abnormality precluding transrectal ultrasound

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of prostate cancer | When histopathology results available, expected to be within 14 days following biopsy
  Absolute differences in PCa detection rate will be calculated with 95% CIs. If lower bound of 97.5% CI for the difference in cancer detection rates of LA TP biopsy compared with TRUS biopsy is greater than -5%, then TP biopsy will be deemed non-inferior. If lower bound is greater than 0, TP will be deemed superior.

SECONDARY OUTCOMES:
Procedure tolerability | Immediately following test
  The pain score of the procedure reported by patient
General health-related quality of life | Baseline and 30 days post-biopsy
  EQ-5D-5L
Quality of life concerning urinary symptoms | Baseline and 30 days post-biopsy
  International Prostate Symptom Score (I-PSS)
Quality of life concerning erectile function | Baseline and 30 days post-biopsy
  International Index of Erectile Function (IIEF)
Rate of procedure induced sepsis | 1 week to 30 days post-biopsy
Detection rates of patients with clinically significant PCa | When histopathology results available, expected to be within 14 days following biopsy
  Ca Prostate with Gleason score larger or equal to 3+4
Maximum cancer core length (MCCL, mm) | When histopathology results available, expected to be within 14 days following biopsy
Proportion of men go on to undergo definitive curative treatment for local disease (including surgery and radiotherapy) | After treatment decision, expected to be within 30 days following biopsy
Procedure times (minutes) | During test
  Time from start of ultrasound probe insertion to probe removal
Cost per diagnosis of cancer (HKD) | 30 days post-biopsy
  The cost of each diagnosis based on the equipment, manpower and medication

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Lam, Principal Investigator — The University of Hong Kong
Locations (1):
- Division of Urology, Department of Surgery, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Hsing AW, Tsao L, Devesa SS. International trends and patterns of prostate cancer incidence and mortality. Int J Cancer. 2000 Jan 1;85(1):60-7. doi: 10.1002/(sici)1097-0215(20000101)85:13.0.co;2-b. PMID 10585584
- [Background] Klotz L. Active surveillance for low-risk prostate cancer. Curr Urol Rep. 2015 Apr;16(4):24. doi: 10.1007/s11934-015-0492-z. PMID 25764118
- [Background] Hodge KK, McNeal JE, Terris MK, Stamey TA. Random systematic versus directed ultrasound guided transrectal core biopsies of the prostate. J Urol. 1989 Jul;142(1):71-4; discussion 74-5. doi: 10.1016/s0022-5347(17)38664-0. PMID 2659827
- [Background] Presti JC Jr, O'Dowd GJ, Miller MC, Mattu R, Veltri RW. Extended peripheral zone biopsy schemes increase cancer detection rates and minimize variance in prostate specific antigen and age related cancer rates: results of a community multi-practice study. J Urol. 2003 Jan;169(1):125-9. doi: 10.1016/S0022-5347(05)64051-7. PMID 12478119
- [Background] Nakai Y, Tanaka N, Anai S, Miyake M, Hori S, Tatsumi Y, Morizawa Y, Fujii T, Konishi N, Fujimoto K. Transperineal template-guided saturation biopsy aimed at sampling one core for each milliliter of prostate volume: 103 cases requiring repeat prostate biopsy. BMC Urol. 2017 Apr 5;17(1):28. doi: 10.1186/s12894-017-0219-1. PMID 28381267
- [Background] Falzarano SM, Zhou M, Hernandez AV, Moussa AS, Jones JS, Magi-Galluzzi C. Can saturation biopsy predict prostate cancer localization in radical prostatectomy specimens: a correlative study and implications for focal therapy. Urology. 2010 Sep;76(3):682-7. doi: 10.1016/j.urology.2009.11.067. Epub 2010 Mar 5. PMID 20206973
- [Background] Tsu JH, Ma WK, Chan WK, Lam BH, To KC, To WK, Ng TK, Liu PL, Cheung FK, Yiu MK. Prevalence and predictive factors of harboring fluoroquinolone-resistant and extended-spectrum beta-lactamase-producing rectal flora in Hong Kong Chinese men undergoing transrectal ultrasound-guided prostate biopsy. Urology. 2015 Jan;85(1):15-21. doi: 10.1016/j.urology.2014.07.078. Epub 2014 Nov 8. PMID 25444632
- [Background] Meyer AR, Joice GA, Schwen ZR, Partin AW, Allaf ME, Gorin MA. Initial Experience Performing In-office Ultrasound-guided Transperineal Prostate Biopsy Under Local Anesthesia Using the PrecisionPoint Transperineal Access System. Urology. 2018 May;115:8-13. doi: 10.1016/j.urology.2018.01.021. Epub 2018 Feb 1. PMID 29409845
- See also: Prostate cancer incidence statistics. Cancer research UK. London, United Kingdom: cancer research 2014. — http://www.cancerresearchuk.org/cancer-info/cancerstats/types/prostate/incidence/#source9
- See also: The Hong Kong cancer registry. Hospital Authority, Hong Kong. — http://www3.ha.org.hk/cancereg/topten.html
- See also: 11. United States Food and Drug Adminstration Approval of PrecisionPoint Transperineal Access System. — http://www.accessdata.fda.gov/cdrh_docs/pdf16/k160414.pdf

DOCUMENTS (1):
  • Study Protocol (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04108871/Prot_000.pdf